CLINICAL TRIAL: NCT03299738
Title: A Phase 1 Study Evaluating Safety and Efficacy of C-CAR011 in Subjects With B-cell Non-Hodgkin Lymphoma (NHL)
Brief Title: A Study Evaluating Safety and Efficacy of C-CAR011 in Subjects With B-NHL
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai AbelZeta Ltd. (Industry)
Collaborators: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBMG-C2017006
Record Dates: First submitted 2017-09-28; First posted 2017-10-03 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Refractory or Relapsed B-cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- C-CAR011 (Experimental): Lymphocytes will be transduced with lentiviral vector containing CAR-CD19 gene
  Interventions: Biological: C-CAR011

INTERVENTIONS:
Biological: C-CAR011 — Autologous 2nd generation CD19-directed CAR-T cells, single infusion intravenously at a target dose of 0.5-5.0 x 10^6 anti-CD19 CAR+ T cells/kg
  Other Names: Anti-CD19 Chimeric Antigen Receptor T cell

SUMMARY:
This is a single arm, single-center, non-randomized study to evaluate the safety and efficacy of C-CAR011 in relapsed or refractory B cell Non-Hodgkin Lymphoma (NHL).

DETAILED DESCRIPTION:
The study will include the following sequential phases: Screening, Pre-Treatment (Cell Product Preparation, Lymphodepleting Chemotherapy), Treatment and Follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteered to participate in this study and signed informed consent
2. Age 18-70 years old, male or female
3. Relapse or refractory B cell non-Hodgkin's lymphoma

   * 1. Histologically diagnosed as DLBCL (including PMBCL) or follicular lymphoma (grade Ⅲb) according to the NCCN non-Hodgkin's lymphoma Clinical Practice Guidelines (2017 Version 1)

     * Progressive disease after the last standard chemotherapy regimens per the IWG Response Criteria (1999)
     * Stable disease after the last standard chemotherapy regimens (at least 4 cycles of first-line therapy or 2 cycles of later-line therapy) per the IWG Response Criteria (1999)
     * Relapse or progressive disease within 12 months after autologous stem cell transplantation (SCT)
   * 2. Follicular lymphoma (stage Ⅲ-Ⅳ) (gradeⅠ-Ⅲa)

     * At least 2 combination chemotherapy regimens (excluding single agent monoclonal antibody)
     * Relapse or progressive disease within 1 year after last chemotherapy regimens
   * 3. Mantle cell lymphoma

     * Relapse after 1st CR or persistent disease, and not eligible or appropriate for SCT
     * Relapse or progressive disease within 1 year after the last chemotherapy regimens
     * Relapse or progressive disease within 12 months after autologous SCT
4. All subjects must have received anti-CD20 monoclonal antibody (unless tumor is CD20-negative) and anthracycline-containing chemotherapy regimens according to NCCN non-Hodgkin lymphoma Clinical Practice Guidelines (2017 Version 1)
5. At least one measurable lesion per revised IWG Response Criteria (the longest diameter of the tumor ≥ 1.5 cm)
6. Expected survival ≥ 12 weeks
7. ECOG score 0-1
8. Left ventricular ejection fraction (LVEF) ≥ 50% (detected by echocardiography)
9. No active pulmonary infections, normal pulmonary function and oxygen saturation ≥ 92% on room air
10. At least 2 weeks from receiving previous treatment (radiotherapy or chemotherapy) prior to leukapheresis, or at least 4 weeks from monoclonal antibody therapy prior to CAR T cell therapy
11. No contraindications of leukapheresis
12. Female subjects in childbearing age, their serum or urine pregnancy test must be negative, and must agree to take effective contraceptive measures during the trial

Exclusion Criteria:

1. History of allergy to cellular products
2. Laboratory tests: absolute neutrophil count < 1.0 × 10^9 /L, platelet count < 50 × 10^9 /L, serum albumin < 30 g/L, serum bilirubin > 1.5 ULN, serum creatinine > ULN, ALT/AST > 3 ULN
3. History of CAR T cell therapy or any other genetically modified T cell therapy
4. Relapse after allogeneic hematopoietic stem cell transplantation
5. Active infections that require treatment (uncomplicated urinary tract infections and bacterial pharyngitis are allowed), prophylactic antibiotic, antiviral and antifungal treatment are permitted
6. Hepatitis B or hepatitis C virus infection (including carriers), syphilis, as well as acquired or congenital immune deficiency diseases, including but not limited to HIV infection
7. Class III or IV heart failure according to the NYHA Heart Failure Classifications
8. QT interval prolongation ≥ 450 ms
9. History of epilepsy or other central nervous system disorders
10. Evidence of CNS lymphoma by head enhancement scan or magnetic resonance imaging
11. History of other primary cancers, with the following exceptions

    * Excisional non-melanoma (e.g. cutaneous basal cell carcinoma)
    * Cured in situ carcinoma (e.g. cervical cancer, bladder cancer, breast cancer)
12. Autoimmune diseases that require treatment, immune deficiency diseases or other diseases that require immunosuppressive therapy
13. Used of systemic steroids within two weeks (using inhaled steroids is an exception)
14. Women who are pregnant or lactating, or who have breeding intent in 6 months
15. Participated in any other clinical trial within three months
16. Any situation that investigators believe the risk of the subjects is increased or results of the trial are disturbed

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-12 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Safety: Vital signs, physical examination, clinical laboratory tests, incidence of adverse events (AEs) and serious adverse events (SAEs) | 12 weeks
  Vital signs, physical examination, clinical laboratory tests, incidence of adverse events (AEs) and serious adverse events (SAEs)
Overall response rate (ORR) | 12 weeks

SECONDARY OUTCOMES:
Overall response rate (ORR) | 6 months
Overall response rate (ORR) | 12 months
Duration of remission (DOR) | 12 months
Progression free survival (PFS) | 12 months
Overall survival (OS) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Huilai Zhang, Principal Investigator — Department of Lymphoma, Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Department of Lymphoma, Tianjin Medical University Cancer Institute and Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: Undecided